CLINICAL TRIAL: NCT02622659
Title: The Efficacy and Safety Study of Fuganlin Oral Liquid in Children With Influenza (Acute Upper Respiratory Infection)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012Pro170EKZY
Record Dates: First submitted 2015-11-16; First posted 2015-12-04 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2015-11

CONDITIONS: Acute Upper Respiratory Infection
Keywords: acute upper respiratory infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fuganlin Oral Liquid (Experimental): Fuganlin Oral Liquid:oral
  less than 1 years old: 5mL each time and three times a day
  1~3 years old: 10mL each time and three times a day
  4~6 years old: 10mL each time and four times a day
  7~12 years old: 10mL each time and five times a day
  Xiaoer Jiebiao Oral Liquid placebo:oral
  1~2 years old: 5mL each time and twice a day
  3~5 years old: 5mL each time and three times a day
  6~14 years old: 10mL each time and twice a day
  Interventions: Drug: Fuganlin Oral Liquid
- Xiaoer Jiebiao Oral Liquid (Active Comparator): Xiaoer Jiebiao Oral Liquid:oral
  1~2 years old: 5mL each time and twice a day
  3~5 years old: 5mL each time and three times a day
  6~14 years old: 10mL each time and twice a day
  Fuganlin Oral Liquid placebo:oral
  less than 1 years old: 5mL each time and three times a day
  1~3 years old: 10mL each time and three times a day
  4~6 years old: 10mL each time and four times a day
  7~12 years old: 10mL each time and five times a day
  Interventions: Drug: Xiaoer Jiebiao Oral Liquid

INTERVENTIONS:
Drug: Fuganlin Oral Liquid — less than 1 years old: 5mL each time and three times a day
  1~3 years old: 10mL each time and three times a day
  4~6 years old: 10mL each time and four times a day
  7~12 years old: 10mL each time and five times a day
  Other Names: No other names
  Arms: Fuganlin Oral Liquid
Drug: Xiaoer Jiebiao Oral Liquid — 1~2 years old: 5mL each time and twice a day
  3~5 years old: 5mL each time and three times a day
  6~14 years old: 10mL each time and twice a day
  Other Names: No other names
  Arms: Xiaoer Jiebiao Oral Liquid

SUMMARY:
Randomized, double blind, double dummy, positive drug parallel comparison, multi-centre clinical trial to assess the efficacy and safety of Fuganlin Oral Liquid in children with influenza (acute upper respiratory infection).

DETAILED DESCRIPTION:
Treatment group: Fuganlin Oral Liquid 10mL. Control group: Xiaoer Jiebiao oral liquid 100mL. Treatment for one week. Patients who were recovered within one week can withdrawal at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as acute upper respiratory infection.
2. Patients with Traditional Chinese Medicine syndrome of qi deficiency and wind-heat.
3. Patients aged 1 to 12 years.
4. With course of disease in 48 hours or less.
5. Signed informed consent by a Parent or legal guardians.

Exclusion Criteria:

1. Patients diagnosed as tonsillitis, bronchitis, bronchiolitis, pneumonia;
2. Patients have a history of hyperpyretic convulsion;
3. Severe malnutrition, rickets patients and merge the heart, brain, liver, kidney and hematopoietic system and other serious primary diseases;
4. The increased of serum creatinine (Cr), blood urea nitrogen (BUN), alanine aminotransferase (ALT), and urinary protein, urine RBC above "+", which can not use the test illness or possibly combined disease conditions to explain;
5. Patients with allergic physique (Allergic to above two kinds of substance), allergic to the composition of the preparation or control drug;
6. According to the doctors' determination,likely to loss to follow up.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 468 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The duration of cold symptoms | Defined as the time from the onset of the cold to the time achieve a cold cure standard，time average 3 to 7 days
  Cold diagnostic criteria：
  1. nasal congestion, runny nose, sneezing, itchy throat, or pain, cough
  2. The chills, fever, no sweat or less sweat, headache, limb sour
  3. The total number normal or low of white blood cells, neutropenia, relative increase in lymphocytes
  Cold cure criteria:
  1. fever, aversion to wind individual symptoms disappeared
  2. nasal congestion, runny nose, sore throat, cough individual symptoms disappeared

CONTACTS AND LOCATIONS:
Overall Officials: Cao xia, MD, Principal Investigator — Chongqing First People's Hospital; Yan yunying, MD, Principal Investigator — Nanning maternal and Child Health Hospital; Hu suping, MD, Principal Investigator — Nanchang City Hospital of integrated traditional Chinese and Western Medicine; Wang leping, MD, Principal Investigator — Changzhou traditional Chinese medicine hospital; Liu Dexing, MD, Principal Investigator — Liuzhou traditional Chinese medicine hospital; Qi Shihe, MD, Principal Investigator — Xiangyang Central Hospital; Ding Lijun, MD, Principal Investigator — Handan traditional Chinese medicine hospital; Yang Liping, MD, Principal Investigator — Changzhi City People's Hospital; Feng Ziwei, MD, Principal Investigator — Luohe traditional Chinese medicine hospital
Locations (1):
- Luohe traditional Chinese medicine hospital, Luohe, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided